CLINICAL TRIAL: NCT01258452
Title: Randomized, Balanced, Single Dose, Cross-Over Study to Evaluate the Effects of Food Ingestion on the Pharmacokinetics of CHF 5074 in Healthy Young Male Subjects
Brief Title: Study to Evaluate the Effects of Food Ingestion on the Pharmacokinetics of CHF 5074 in Healthy Young Male Subjects
Acronym: CT03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CERESPIR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-1013-PR-0052
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 1-(3',4'-dichloro-2-fluoro(1,1'-biphenyl)-4-yl)cyclopropanecarboxylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF 5074 (fed group) (Experimental): oral tablet, single dose
  Interventions: Drug: CHF 5974
- CHF 5074 (fasting group) (Experimental): oral tablet, single dose
  Interventions: Drug: CHF 5074

INTERVENTIONS:
Drug: CHF 5074 — Drug is administered to subject in a fasting state
  Arms: CHF 5074 (fasting group)
Drug: CHF 5974 — Drug is administered to subject after consumption of a high fat, high calorie meal
  Arms: CHF 5074 (fed group)

SUMMARY:
To evaluate the effects of a high-calorie high-fat meal on the extent and rate of absorption of CHF 5074 after single oral administration in young healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is judged to be in good health on the basis of medical history, complete physical examination including vital signs, 12-lead electrocardiogram (ECG) and standard laboratory tests.
* Subject has a body mass index between 18 and 30 kg/m^2, inclusive.

Exclusion Criteria:

* Medical history (within the last 10 years) of major cardiovascular, hepatic or renal disease.
* Abnormal result of liver function tests, renal function tests or thyroid tests performed at screening.
* Significant allergic conditions that require medical treatment
* Use of any psychoactive, recreational or prescription drug within the 4 weeks prior to study drug administration.
* Use of ibuprofen, sulindac sulfide, indomethacin, flurbiprofen within 2 weeks prior to study drug administration.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
area under the curve of plasma CHF 5074 levels from 0 to 96 hours (AUC 0-96) | from Day 1 to Day 5
peak CHF 5074 plasma concentration (Cmax) | from Day 1 to Day 5

SECONDARY OUTCOMES:
the time of occurrence of Cmax (Tmax) | from Day 1 to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Magdy L. Shenouda, MD, Principal Investigator — Iberica Clinical Research Center
Locations (1):
- Iberica Clinical Research Center, Eatontown, New Jersey, United States